CLINICAL TRIAL: NCT06369909
Title: Study on AI-assisted Multimodal Diagnosis System of Autoimmune Pancreatitis Based on the Mechanism of Tfh Activation by Intestinal Bacteria and Endosonographic Features
Brief Title: Study on AI-assisted Multimodal Diagnosis System of Autoimmune Pancreatitis
Status: Recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Tianjin Medical University General Hospital (Other); The Second Hospital of Hebei Medical University (Other)
Responsible Party: Principal Investigator, Wu Xi, Professor, Peking Union Medical College Hospital
Other Study IDs: K5507
Record Dates: First submitted 2024-04-06; First posted 2024-04-17 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-04

CONDITIONS: Autoimmune Pancreatitis
Keywords: Autoimmune pancreatitis; Endoscopic ultrasonography; Artificial intelligence; Follicular helper T cells; Klebsiella pneumoniae
MeSH Terms: conditions — Autoimmune Pancreatitis | interventions — Endoscopic Ultrasound-Guided Fine Needle Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — 10 mL of peripheral blood sample, stool sample, fine needle biopsy samples of pancreatic lesions in autoimmune pancreatitis, biopsy samples of duodenal mucosa.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- AIP group: Suspected AIP, pancreatic mass patients who have not initiated steroid hormone therapy
  Interventions: Procedure: EUS-FNA
- Control group: Pancreatic mass patients considering malignancy and planning to undergo EUS-FNA
  Interventions: Procedure: EUS-FNA

INTERVENTIONS:
Procedure: EUS-FNA — For patients with pancreatic masses, EUS-FNA is performed to confirm pathological diagnosis, and pancreatic biopsy samples and duodenal mucosal biopsy samples are collected.

SUMMARY:
The existing comprehensive diagnostic system for autoimmune pancreatitis (AIP) is complex, with multidimensional clinical information including morphological changes and a lack of specific biomarkers. Endoscopic ultrasound (EUS) can provide all the elements for morphological diagnosis of AIP, but the long learning curve and large observer differences make it difficult to popularize and promote. The cooperation units of the three regions in this project have found in the early stage that Klebsiella pneumoniae (KP) induced follicular helper T cells (Tfh) activation is an important mechanism of AIP, but the identification of pathogenic components of the strain and clinical validation need to be explored. We have established a national multicenter AIP queue in the early stage and extracted EUS audio-visual features to establish a scoring model, but intelligent assistance is still needed to improve efficiency. Therefore, we plan to integrate gut microbiota, Tfh activation markers, and EUS imaging features to establish an AI assisted multimodal diagnostic system for AIP. This study will collaborate across multiple centers to identify and validate the components that induce Tfh activation in KP bacterial cells, to extract EUS pancreatic ultrasound features and optimize artificial intelligence assisted diagnostic algorithms, and to establish and validate an artificial intelligence assisted multimodal diagnostic system based on clinical information, biomarkers, and EUS. The aim of this study is to provide new diagnosis and treatment evaluation methods for AIP with high accuracy, convenience, and easy promotion for clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* From the beginning of the study to the end of the study, patients with pancreatic solid lesions suspected or diagnosed with AIP were treated at Peking Union Medical College Hospital and related research centers.
* The patients themselves and their families understood and were willing to participate in this study, and signed an informed consent form.
* The diagnosis of AIP must comply with the criteria of the Chinese Guidelines for the Diagnosis and Treatment of Autoimmune Pancreatitis (2022).

Exclusion Criteria:

* Individuals who are not suitable for endoscopic examination, including but not limited to: generally poor condition, severe cardiovascular and pulmonary diseases, and difficulty tolerating the examination, coagulation disorders and those who are deemed unsuitable for endoscopic examination by an endoscopist after a face-to-face consultation.
* Patients or family members are unable to understand the conditions and objectives of this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with pancreatic solid lesions suspected or diagnosed with AIP. The diagnosis of AIP must comply with the criteria of the Chinese Guidelines for the Diagnosis and Treatment of Autoimmune Pancreatitis (2022).
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2024-01-31 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Tfh level in blood | from enrollment to 3 years
  The type and level of follicular helper T cells in peripheral blood for each patient
Microbiota composition measured by 16S rRNA sequencing | from enrollment to 3 years
  The gut microbiota of fecal samples and the intestinal microbiota of duodenal biopsy samples using 16S rRNA sequencing for each patient
AI-EUS differentiation | from enrollment to 3 years
  The differentiation of EUS graphs by AI system
Cytokine level in blood | from enrollment to 3 years
  IL-4、IL-21、CXCL13、IgG、IgE level in peripheral blood
Single cell sequencing | At the time of enrollment
  Single cell sequencing results of pancreatic lesion biopsy samples and duodenal mucosal biopsy samples in autoimmune pancreatitis.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China